CLINICAL TRIAL: NCT01488058
Title: A Randomised Controlled Trial Comparing Internet Based Cognitive Behavioural Therapy for Major Depressive Disorder Plus a Cognitive Bias Modification Intervention (OxIGen) vs. Internet Based Cognitive Behavioural Therapy for Major Depressive Disorder vs. a Waitlist Control on Symptoms of Depression and Negative Interpretation Bias.
Brief Title: Cognitive Bias Modification (CBM) and Internet Cognitive Behavioural Therapy (iCBT) for Depression- A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alishia Williams (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor-Investigator, Alishia Williams, Principal Investigator, St Vincent's Hospital
Organization: St Vincent's Hospital, Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/055; ACTRN12611001221943 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Other): Waitlist control
  Interventions: Other: Waitlist Control
- Group 1 (Experimental): CBM intervention (OxIGen) plus Internet based Cognitive Behavioural Therapy for depression
  Interventions: Other: OxIGen + iCBT

INTERVENTIONS:
Other: OxIGen + iCBT — OxIGen is an Internet-based intervention taking place over 1 week followed by iCBT, an Internet-based treatment for depression taking place over 10 weeks.
  Arms: Group 1
Other: Waitlist Control — Waitlist will receive iCBT at week 11
  Arms: Group 2

SUMMARY:
Cognitive accounts of depression and anxiety emphasize the importance of cognitive biases in the maintenance of disorders. One specific bias is the interpretation of ambiguous information. A negative interpretation bias is defined as a systematic tendency to interpret potentially ambiguous information in a negative rather than benign way and this bias has been associated with symptoms of depression. Research has led to the recent development of computerized cognitive bias modification (CBM) techniques to augment such biases and it has been suggested that CBM techniques may be useful as an adjunct to current treatments to enhance maintenance of treatment gains and minimize relapse rates. The fact that CBM procedures lend themselves to being delivered remotely, are cost-effective, and can be self-paced in ways that suit the patient make them an ideal candidate for inclusion in the Internet-based cognitive behavioural therapy (iCBT) programs currently offered through St. Vincent's Hospital and the University of New South Wales. Therefore, the primary aim of the current trial is to evaluate the acceptability and effectiveness of adding CBM procedures to the existing iCBT modules offered through St. Vincent's Hospital and the University of New South Wales. It is expected that iCBT + CBM will result in superior treatment outcomes as indexed by a standardized clinical battery.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of the American Psychiatric Association - 4th edition (DSM-IV) criteria for Major Depressive Disorder,
* Internet access + printer access,
* Australian resident,
* Fluent in written and spoken English.

Exclusion Criteria:

* Current substance abuse/dependence,
* Psychotic mental illness (Bipolar or Schizophrenia),
* Current or planned psychological treatment during study duration,
* Change in medication during last 1 month or intended change during study duration,
* Use of Benzodiazepines,
* Suicidal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in score on the Beck Depression Inventory - second edition (BDI-II). | Administered at baseline, post-intervention (1 week), and post treatment (iCBT; 11 weeks)

SECONDARY OUTCOMES:
Change on the Scrambled Sentences Task (SST)- electronic version. | Administered at baseline, post-intervention (1 week).
Change on Prospective Imagery Test (PIT). | Administered at baseline, post-intervention (1 week).
Change on the Kessler-10 (K10). | Administered at baseline, before each iCBT lesson, and post-treatment (week 11).
Change on WHO Disability Assessment Scale (WHO-DAS). | Administered baseline and post-treatment (iCBT; 11 weeks).
Change on the Repetitive Thinking Questionnaire (RTQ). | Administered at baseline, post intervention (week 1), and post-treatment (iCBT; 11 weeks).
Change on the State Trait Anxiety Inventory (STAI). | Administered at baseline, post intervention (week 1), and post-treatment (iCBT; 11 weeks).
Change on the Ambiguous Sentence Task (AST). | Administered at baseline and post-intervention (week 1).
Change in score on the Patient Health Questionnaire-9 (PHQ-9). | Administered at baseline, post intervention (week 1), and post treatment (week 11).

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Andrews, AO, MD, Principal Investigator — St. Vincent's Hospital, The University of New South Wales; Alishia Williams, PhD; MPsychol(Clinical), Principal Investigator — St. Vincent's Hospital, The University of New South Wales
Locations (1):
- St. Vincent's Hospital, Darlinghurst, New South Wales, Australia